CLINICAL TRIAL: NCT06053866
Title: Prevalence of Erthropoietin Stimulating Agents Hyporesponsiveness and Its Correlation With Cardiovascular Morbidities in Hemodialysis Patients in Assiut University Hospital
Brief Title: Prevalence of Erythropoiesis Stimulating Agents Hyporesponsiveness in Dialysis Patients in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Feby Rasmy Khalifa Makar, Doctor, Assiut University
Other Study IDs: Erythropoietin resistance
Record Dates: First submitted 2023-09-13; First posted 2023-09-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Erythropoietin Resistant Anemia (EPO Resistant Anemia)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* The prevalence of erthropoietin stimulating agents hyporesponsiveness in hemodialysis patients in Assiut university hospital
* Assessment of cardiovascular diseases risk in patients with erythropoiesis stimulating agents hyporesponsiveness in hemodialysis patients in Assiut university hospital

DETAILED DESCRIPTION:
Anemia is common in patients with chronic kidney disease. The routine use of erthropoietin in anemia control has reduced morbidity and mortality rates in patients with chronic kidney disease. Despite an increase in the use and average dose of recombinant human epoetin over the last 15 years, a substantial percentage of patients still don't achieve hemoglobin targets recommend by international guidelines. The definition of recombinant human epoetin resistance has been introduced to identify those patients in whom the target hemoglobin level is not attained despite a greater than usual dose of erthropoietin stimulating agent. In recent years, increasing attention has been paid to the relationship between dialysis, increased inflammatory stimulus, malnutrition, and erythropoiesis stimulating agents response. Erythropoiesis stimulating agents hyporesponsiveness was defined by the erythropoietin resistance index, which was the erythropoietin dose per week divided by body weight and Hemoglobin level . The resistance to erythropoiesis stimulating agents is directly related with incident comorbidity in patients on hemodialysis and it can be interpreted as a useful marker of early mortality. Patients with higher erythropoietin resistance index values had a higher all cause mortality rate and cardiovascular mortality rate. Erythropoietin resistance index was related with left ventricular mass index, left ventricle systolic function and cardiovascular events in patients with hemodialysis. By monitoring of erthropoietin resistance index, early identification of the epoetin resistance may be useful to predict the cardiovascular risk in hemodialysis patients

ELIGIBILITY:
Inclusion Criteria:

* age more than 18
* End stage renal disease patients undergoing regular hemodialysis in Assiut University Hospital - Hemodialysis unit for duration at least 3 months

Exclusion Criteria:

* acute infectious disease within one month
* active liver disease or cancer
* recent blood transfusion or surgical intervention
* active bleeding or hemorrhage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: End stage renal disease patients undergoing regular hemodialysis for at least 3 months duration
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prevalence of Erythropoiesis stimulating agents hyporesponsiveness in dialysis patients in Assiut university hospital | One year
  Erythropoiesis resistance index which is the erythropoietin dose per week divided by body weight and Hemoglobin level

SECONDARY OUTCOMES:
Assessment of cardiovascular diseases risk in hemodialysis patients with erythropoiesis stimulating agents hyporesponsiveness | One year
  Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Hewida Abdelhakem Nafady, Principal Investigator — Assiut University; Radwa Awad abdelhafez, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Lurdes Agostinho Cabrita A, Pinho A, Malho A, Morgado E, Faisca M, Carrasqueira H, Silva AP, Neves PL. Risk factors for high erythropoiesis stimulating agent resistance index in pre-dialysis chronic kidney disease patients, stages 4 and 5. Int Urol Nephrol. 2011 Sep;43(3):835-40. doi: 10.1007/s11255-010-9805-9. Epub 2010 Jul 17. PMID 20640598
- [Background] Bamgbola OF, Kaskel FJ, Coco M. Analyses of age, gender and other risk factors of erythropoietin resistance in pediatric and adult dialysis cohorts. Pediatr Nephrol. 2009 Mar;24(3):571-9. doi: 10.1007/s00467-008-0954-3. Epub 2008 Sep 18. PMID 18800231
- [Background] Del Vecchio L, Pozzoni P, Andrulli S, Locatelli F. Inflammation and resistance to treatment with recombinant human erythropoietin. J Ren Nutr. 2005 Jan;15(1):137-41. doi: 10.1053/j.jrn.2004.09.024. PMID 15648023
- [Background] Tanaka S, Kitamura H, Tsuruya K, Kitazono T, Nakano T; FKR Study Collaboration Group. Prevalence, treatment status, and predictors of anemia and erythropoietin hyporesponsiveness in Japanese patients with non-dialysis-dependent chronic kidney disease: a cross-sectional study. Clin Exp Nephrol. 2022 Sep;26(9):867-879. doi: 10.1007/s10157-022-02227-8. Epub 2022 May 4. PMID 35507237
- [Background] Okazaki M, Komatsu M, Kawaguchi H, Tsuchiya K, Nitta K. Erythropoietin resistance index and the all-cause mortality of chronic hemodialysis patients. Blood Purif. 2014;37(2):106-12. doi: 10.1159/000358215. Epub 2014 Mar 5. PMID 24603656
- [Background] Lopez-Gomez JM, Portoles JM, Aljama P. Factors that condition the response to erythropoietin in patients on hemodialysis and their relation to mortality. Kidney Int Suppl. 2008 Dec;(111):S75-81. doi: 10.1038/ki.2008.523. PMID 19034333
- [Background] Lu X, Zhang J, Wang S, Yu Q, Li H. High Erythropoiesis Resistance Index Is a Significant Predictor of Cardiovascular and All-Cause Mortality in Chinese Maintenance Hemodialysis Patients. Mediators Inflamm. 2020 Nov 26;2020:1027230. doi: 10.1155/2020/1027230. eCollection 2020. PMID 33293895
- [Background] Chung S, Song HC, Shin SJ, Ihm SH, Park CS, Kim HY, Yang CW, Kim YS, Choi EJ, Kim YK. Relationship between erythropoietin resistance index and left ventricular mass and function and cardiovascular events in patients on chronic hemodialysis. Hemodial Int. 2012 Apr;16(2):181-7. doi: 10.1111/j.1542-4758.2011.00644.x. PMID 22103889